CLINICAL TRIAL: NCT03427073
Title: A Phase I Open-label Multicentre Dose-escalation Study of Subcutaneous ALM201 in Patients With Advanced Ovarian Cancer and Other Solid Tumours
Brief Title: A Phase I Dose-escalation Study of Subcutaneous ALM201 in Patients With Advanced Ovarian Cancer and Other Solid Tumours
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: to re-evaluate biomarker strategy for recruitment to Part 2
Sponsor: Almac Discovery (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALM201/0001
Record Dates: First submitted 2015-03-05; First posted 2018-02-09 (Actual); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Solid Tumors; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solid tumours (Experimental): Part 1 - Dose-escalation of ALM201 in patients with advanced solid tumours
  Daily dosing of ALM201 on Days 1-5, 8-12 and 15-19 of 21 day cycle. Escalating dose cohorts
  Interventions: Drug: ALM201
- Ovarian cancer (Experimental): Part 2 - Dose-expansion of ALM201 Maximum Tolerated Dose (MTD) in patients with advanced ovarian cancer
  Daily dosing of ALM201 on Days 1-5, 8-12 and 15-19 of 21 day cycle at the MTD determined in Part 1
  Interventions: Drug: ALM201

INTERVENTIONS:
Drug: ALM201 — Drug: ALM201 administered subcutaneously

SUMMARY:
ALM201/0001 is a Phase I, open-label, dose-escalation study of the safety, tolerability and pharmacokinetics (PK) of ALM201.

Part 1 will be a dose-escalation study. Patients with advanced solid tumours will receive daily doses of ALM201 on Days 1-5, 8-12 and 15-19 in 21 day cycles.

Part 2 will be a dose-expansion of the Maximum Tolerated Dose (MTD) determined in Part 1. Patients with advanced ovarian cancer will be enrolled with the main objective to determine the recommended Phase II dose.

DETAILED DESCRIPTION:
ALM201 is a peptide with anti-angiogenic activity in a range of in-vitro and ex-vivo models. ALM201/0001 is a Phase I, multicentre, open-label, dose-escalation study of the safety, tolerability and pharmacokinetics (PK) of ALM201. The study is divided into two parts.

Part 1 will enrol patients with advanced solid tumours. Patients will receive subcutaneous injection of ALM201 on Days 1-5, 8-12 and 15-19 in 21 day cycles. Patients can receive up to 8 cycles of treatment. Enrolment will follow an accelerated dose-escalation schedule until grade 2 drug-related adverse events are observed, at this point the 3+3 enrolment design will be used. There will be at least 1 week stagger between the first and subsequent patients in a new cohort dose. Dose increments will not exceed 100% escalation and will be guided by data generated from previous cycles. The dose and possibly the schedule will be adjusted to determine the Maximum Tolerated Dose (MTD).

Part 2 will enrol patients with advanced ovarian cancer whose tumour has a proangiogenic profile as assessed by an angiogenesis gene signature biomarker. Patients will receive ALM201 at a dose and schedule established in Part 1.

Patients will undergo safety and tumour assessments as well as blood draws for PK profiling. The safety assessments will involve physical examination, vital signs, biochemistry and haematology laboratory screens as well as immunogenicity testing. Tumour assessments will involve computed tomography (CT) or magnetic resonance imaging (MRI) scans at screening and after every 2 cycles during cycles 1 -8. Patients will be asked to provide consent for access to archived tumour tissue and for fresh biopsies to be taken at pre-dose, tumour response and/or point of disease progression for potential biomarker and pharmacodynamic assessments. PK profiling will be carried out in Cycles 1, 2, 4, 6 and 8.

ELIGIBILITY:
Inclusion Criteria:

* Part 1 Specific Inclusion Criterion

  *Patients with histologically and/or cytologically confirmed advanced solid tumour for whom no standard effective therapy is available or felt likely to be of limited efficacy and in whom a rationale for use of an anti-angiogenic treatment approach exists. Note: Previous use of anti-angiogenic therapy is allowed if tolerated
* Part 2 Specific Inclusion Criterion

  *Patients with advanced ovarian cancer, who are intolerant of or whose tumour is resistant to platinums and who have failed to respond to, or have relapsed following, standard therapy and whose tumour has a proangiogenic profile as assessed by the angiogenesis gene signature test. Note: Previous use of anti-angiogenic therapy is allowed if tolerated.
* General Inclusion Criteria for all Patients

  * Measurable or evaluable disease.
  * Recovery from previous treatment to baseline or CTCAE ≤ Grade 1, as determined by CTCAE v4.03 criteria (Appendix B), of reversible toxicities related to prior treatment, with the exception of alopecia, lymphopenia, other non-clinically significant adverse events; recovery from previous radiotherapy other than residual cutaneous effects or stable < Grade 2 gastrointestinal toxicity; complete recovery from surgery other than stable < Grade 2 toxicity.
  * ECOG Performance Status (PS) of 0 or 1.
  * Acceptable haematological, renal and hepatic
  * Women must have either a negative pregnancy test prior to first study drug administration or be post menopausal. Male and female patients of childbearing potential must use appropriate methods birth control.
  * Patients must give written informed consent and understand the requirements of the study

Exclusion Criteria:

For all Patients

* History of inability to tolerate anti-angiogenic therapies e.g. increased blood pressure (BP), proteinuria, prior thromboembolic events.
* Previous history of bowel obstruction, clinical evidence of gastro-intestinal obstruction, large burden of peritoneal disease or evidence of bowel involvement on computed tomography.
* Patents has received:

  * any chemotherapy regimens (including investigational agents) with delayed toxicity within 4 weeks (6 weeks for prior nitrosourea or mitomycin C) of Cycle 1, Day 1, or received chemotherapy regimens given continuously or on a weekly basis which have limited potential for delayed toxicity within 2 weeks of Cycle 1, Day 1.
  * radiotherapy, immunotherapy or biological agents (includes investigational agents) within 4 weeks of Cycle 1, Day 1. Localised palliative radiotherapy is permitted for symptom control.
* Documented, symptomatic or uncontrolled intracranial metastases or primary intracerebral tumours.
* Cancer with leptomeningeal involvement.
* On therapeutic anti-coagulation (aspirin dosing ≤100 mg per oral (PO) daily allowed).
* Previous malignancy, except for non-basal-cell carcinoma of skin or carcinoma-in-situ of the uterine cervix, unless the tumour was treated with curative intent more than 2 years prior to study entry.
* Active cardiac condition or history of significant cardiac condition. Known human immunodeficiency virus positivity.
* Active hepatitis B or C or other active liver disease (other than malignancy).
* Any active, clinically significant, viral, bacterial, or systemic fungal infection within 4 weeks prior to Cycle 1, Day 1.
* Any evidence of severe or uncontrolled systemic conditions or any other issues which make it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Wilson, Professor, Principal Investigator — Centre for Cancer Research and Cell Biology, Queen's University Belfast
Locations (3):
- United Kingdom (3):
  - Centre for Cancer Research and Cell Biology, Queen's University Belfast, Belfast, County Antrim
  - Dept Medical Oncology, The Christie NHS Foundation Trust, Manchester, Lancashire
  - Freeman Hospital, Northern Centre for Cancer Care, Sir Bobby Robson Cancer Trial research Centre, Newcastle, Northumberland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was carried out in three study sites in Belfast, Manchester and Newcastle, UK starting on 27 April 2015.
Pre-assignment Details: Part 1 enrolled adult patients with advanced solid tumours in whom treatment with an anti-angiogenic agent was appropriate. Participants had screening evaluations between Day -1 and -28 before entering the first 21-day treatment cycle.
Groups:
- Cohort 1 - ALM201: One patient received 10 mg IMP from cycle 1 through cycle 6.
- Cohort 2 - ALM201: One patient received 20 mg IMP in cycle 1 and cycle 2.
- Cohort 3 - ALM201: One patient received 40 mg IMP from cycle 1 through cycle 3.
- Cohort 4 - ALM201: Three patients received 80 mg IMP (3 patients during cycle 1, 2 patients in cycle 1 and cycle 2).
- Cohort 5 - ALM201: Three patients received 160 mg of IMP in cycles 1 and 2.
- Cohort 6 - ALM201: Four patients received 200 mg IMP in cycle 1; 3 patients in cycle 1 and 2, 2 patients in cycle 1 through 4 and one patient in cycle 1 through 5.
- Cohort 7 - ALM201: Three patients received 300 mg IMP in cycle 1 and 2; one of them received the IMP in cycle 1 through cycle 6.
- Cohort 8 - ALM201: Four patients received 100 mg IMP in cycle 1; two of them completed cycle 2.
Period: Overall Study
Arm/Group | Cohort 1 - ALM201 | Cohort 2 - ALM201 | Cohort 3 - ALM201 | Cohort 4 - ALM201 | Cohort 5 - ALM201 | Cohort 6 - ALM201 | Cohort 7 - ALM201 | Cohort 8 - ALM201
Started | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 4
Not completed — Disease Progression | 1 | 1 | 1 | 3 | 3 | 4 | 2 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Part 1 enrolled adult patients with advanced solid tumours in whom treatment with an anti-angiogenic agent was appropriate. Participants had screening evaluations between Day -1 and -28 before entering the first 21-day treatment cycle.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - ALM201 | Cohort 2 - ALM201 | Cohort 3 - ALM201 | Cohort 4 - ALM201 | Cohort 5 - ALM201 | Cohort 6 - ALM201 | Cohort 7 - ALM201 | Cohort 8 - ALM201 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 4 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 2 | 2 | 2 | 3 | 2 | 14
  >=65 years | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 2 | 2 | 1 | 1 | 3 | 12
  Male | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 4 | 20
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability - Evaluation of AEs and DLT
Description: All events and suspected dose limiting toxicities (DLTs) were graded according to the CTCAE, version 4.03. A DLT was defined as a Grade 3 or 4 AE that, in the opinion of the CRC, was likely to be related to ALM201 and represented a clinically significant hazard to the patient. Qualifying DLT events were considered to be clinically relevant; e.g. in duration, apparent reversibility, required management, and upon consideration of the patient's medical history and/or concomitant medications. DLT events were also evaluated in terms of what was considered to be an appropriate next escalation step: In the case where the CRC agreed that an escalation step of approximately 33% or lower was merited; the toxicity of concern could be declared a DLT.
  In order to be evaluable for DLT assessment, a patient had to receive at least 80% of their scheduled doses (e.g. 12 of the 15), unless this lack of compliance was due to ALM201-related toxicity.
Time Frame: Adverse event evaluation was done during treatment and follow-up. DLT evaluation was done during cycle 1
Population: Reporting group
Measure: Number; unit: participants
Arm/Group | Cohort 1 - ALM201 | Cohort 2 - ALM201 | Cohort 3 - ALM201 | Cohort 4 - ALM201 | Cohort 5 - ALM201 | Cohort 6 - ALM201 | Cohort 7 - ALM201 | Cohort 8 - ALM201
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 4
participants
  TEAE treatment related | 1 | 0 | 1 | 3 | 3 | 4 | 3 | 4
  TEAE DLT | 1 | 0 | 1 | 1 | 3 | 4 | 3 | 2
  SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  treatment related SAE | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 1

2. Secondary Outcome: Tumour Response Assessment - Best Overall Response
Description: As this was a Phase 1 study, the extent of efficacy data was expected to be limited. Using RECIST Version 1.1, a summary of clinical benefit from patients with evaluable disease was generated via CT scans: Complete Response (CR) = Disappearance of all target & non-target lesions + normalization of tumor marker; Partial Response (PR) ≥ 30% decrease in the sum of LD of target lesions; Progressive Disease (PD) ≥ 20% increase (& 5mm absolute increase) in sum of LD of target lesions or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions; Stable Disease (SD) = Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD or persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits.
Time Frame: Response assessments were done to assess clinical benefit in the efficacy population overall and at the end of cycles 2, 4 and 6, as applicable
Population: Reporting group
Measure: Number; unit: participants
Arm/Group | Cohort 1 - ALM201 | Cohort 2 - ALM201 | Cohort 3 - ALM201 | Cohort 4 - ALM201 | Cohort 5 - ALM201 | Cohort 6 - ALM201 | Cohort 7 - ALM201 | Cohort 8 - ALM201
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 4
participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Overall Response Rate (CR+PR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease (SD) | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 1
  Disease Control Rate (CR+PR+SD) | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 1
  Progressive Disease | 0 | 1 | 0 | 3 | 3 | 1 | 1 | 3
  Not Evaluable (NE+NA) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

3. Secondary Outcome: Pharmacokinetics: Tmax
Description: Tmax was derived from the individual patient plasma concentration versus time profiles of ALM201.
Time Frame: Tmax was determined in cycles 1, 2, 4 and 6 of treatment
Population: Reporting group
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1 - ALM201 | Cohort 2 - ALM201 | Cohort 3 - ALM201 | Cohort 4 - ALM201 | Cohort 5 - ALM201 | Cohort 6 - ALM201 | Cohort 7 - ALM201 | Cohort 8 - ALM201
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 4
hour
  Cycle 1 - Day 1 | 1.45 [1.45 to 1.45] | 1.50 [1.50 to 1.50] | 1.63 [1.63 to 1.63] | 1.53 [0.75 to 2.00] | 1.52 [0.80 to 3.07] | 2.50 [1.50 to 3.08] | 2.00 [0.75 to 4.00] | 1.50 [1.30 to 1.50]
  Cycle 1 - Day 3 | 0.50 [0.50 to 0.50] | 1.00 [1.00 to 1.00] | 1.50 [1.50 to 1.50] | 1.50 [1.05 to 2.00] | 1.52 [1.52 to 2.05] | 2.00 [1.48 to 2.00] | 1.02 [1.00 to 2.00] | 1.61 [0.50 to 2.02]
  Cycle 1 - Day 18: number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 3 | 3 | 2
  Cycle 1 - Day 18 | 1.58 [1.58 to 1.58] | 1.02 [1.02 to 1.02] | 1.00 [1.00 to 1.00] | 1.23 [0.47 to 2.00] | 1.50 [0.50 to 2.00] | 2.03 [1.00 to 3.50] | 1.50 [1.00 to 2.07] | 1.90 [1.45 to 2.35]
  Cycle 2 - Day 18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 2 | 3 | 1
  Cycle 2 - Day 18 | 2.00 [2.00 to 2.00] | 1.00 [1.00 to 1.00] | 1.03 [1.03 to 1.03] | 3.50 [3.50 to 3.50] | 2.00 [2.00 to 2.00] | 1.54 [1.50 to 1.58] | 2.00 [1.48 to 2.13] | 1.02 [1.02 to 1.02]
  Cycle 4 - Day 18: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
  Cycle 4 - Day 18 | 1.53 [1.53 to 1.53] |  |  |  |  | 1.57 [1.00 to 2.13] | 1.12 [1.12 to 1.12] |
  Cycle 6 - Day 18: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 6 - Day 18 | 1.85 [1.85 to 1.85] |  |  |  |  |  | 2.02 [2.02 to 2.02] |

4. Secondary Outcome: Pharmacokinetics: AUC 0-t
Description: AUC 0-t was derived from the individual patient plasma concentration versus time profiles of ALM201.
Time Frame: AUC 0-t was determined in cycles 1, 2, 4 and 6 of treatment
Population: Reporting group
Measure: Geometric Mean (Full Range); unit: ng*h/mL
Arm/Group | Cohort 1 - ALM201 | Cohort 2 - ALM201 | Cohort 3 - ALM201 | Cohort 4 - ALM201 | Cohort 5 - ALM201 | Cohort 6 - ALM201 | Cohort 7 - ALM201 | Cohort 8 - ALM201
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 4
ng*h/mL
  Cycle 1 - Day 1 | 485 [485 to 485] | 1040 [1040 to 1040] | 1920 [1920 to 1920] | 3380 [3100 to 3790] | 6510 [5600 to 7560] | 5860 [3460 to 10200] | 11900 [9470 to 15100] | 6280 [1140 to 14800]
  Cycle 1 - Day 3 | 868 [868 to 868] | 1160 [1160 to 1160] | 898 [898 to 898] | 2970 [2660 to 3430] | 5100 [4970 to 5280] | 6630 [4460 to 11900] | 12500 [10500 to 14700] | 8870 [5380 to 12800]
  Cycle 1 - Day 18: number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 3 | 3 | 2
  Cycle 1 - Day 18 | 817 [817 to 817] | 718 [718 to 718] | 1840 [1840 to 1840] | 3500 [3440 to 3570] | 4930 [4400 to 5400] | 5570 [3900 to 10000] | 12100 [11400 to 12900] | 8100 [7000 to 9370]
  Cycle 2 - Day 18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 2 | 3 | 1
  Cycle 2 - Day 18 | 702 [702 to 702] | 1020 [1020 to 1020] | 1950 [1950 to 1950] | 3230 [3230 to 3230] | 5710 [5710 to 5710] | 5680 [3810 to 8480] | 10400 [7290 to 16700] | 5930 [5930 to 5930]
  Cycle 4 - Day 18: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
  Cycle 4 - Day 18 | 476 [476 to 476] |  |  |  |  | 6110 [4150 to 9010] | 8600 [8600 to 8600] |
  Cycle 6 - Day 18: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 6 - Day 18 | 1040 [1040 to 1040] |  |  |  |  |  | 26700 [26700 to 26700] |

5. Secondary Outcome: Pharmacokinetics: Cmax
Description: Cmax was derived from the individual patient plasma concentration of ALM201.
Time Frame: Cmax of ALM201 following subcutaneous (SC) administration of ALM201 was determined in cycles 1, 2, 4 and 6 of treatment
Population: Reporting group
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Cohort 1 - ALM201 | Cohort 2 - ALM201 | Cohort 3 - ALM201 | Cohort 4 - ALM201 | Cohort 5 - ALM201 | Cohort 6 - ALM201 | Cohort 7 - ALM201 | Cohort 8 - ALM201
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 3 | 4 | 3 | 4
ng/mL
  Cycle 1 - Day 1 | 200 [200 to 200] | 542 [542 to 542] | 592 [592 to 592] | 835 [749 to 892] | 1990 [1730 to 2190] | 1490 [890 to 2690] | 2550 [2100 to 3650] | 1810 [465 to 4600]
  Cycle 1 - Day 3 | 406 [406 to 406] | 614 [614 to 614] | 759 [759 to 759] | 861 [762 to 1090] | 1490 [1390 to 1660] | 1620 [1160 to 3100] | 2690 [2300 to 3260] | 2750 [1450 to 4280]
  Cycle 1 - Day 18: number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 3 | 3 | 2
  Cycle 1 - Day 18 | 352 [352 to 352] | 319 [319 to 319] | 405 [405 to 405] | 1090 [1090 to 1100] | 1350 [1240 to 1420] | 1670 [1230 to 2880] | 2880 [2420 to 3450] | 2330 [2140 to 2530]
  Cycle 2 - Day 18: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 2 | 3 | 1
  Cycle 2 - Day 18 | 288 [288 to 288] | 394 [394 to 394] | 583 [583 to 583] | 849 [849 to 849] | 1870 [1870 to 1870] | 1890 [1280 to 2790] | 2780 [2110 to 4310] | 1790 [1790 to 1790]
  Cycle 4 - Day 18: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
  Cycle 4 - Day 18 | 193 [193 to 193] |  |  |  |  | 1680 [1100 to 2580] | 2140 [2140 to 2140] |
  Cycle 6 - Day 18: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 6 - Day 18 | 470 [470 to 470] |  |  |  |  |  | 6830 [6830 to 6830] |

ADVERSE EVENTS:
Time Frame: AEs were collected from the patient's first dose of IMP, throughout the study until the 30-day follow-up visit. SAEs were followed until considered resolved, returned to baseline, chronically ongoing or otherwise explained by the Principal Investigator.
Description: During the study, AEs were spontaneously reported or elicited during open-ended questioning, examination or evaluation of a patient. Progression of the disease under study was not captured as an AE.
Arm/Group | Cohort 1 - ALM201 | Cohort 2 - ALM201 | Cohort 3 - ALM201 | Cohort 4 - ALM201 | Cohort 5 - ALM201 | Cohort 6 - ALM201 | Cohort 7 - ALM201 | Cohort 8 - ALM201
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/3 | 0/3 | 0/4 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 0/1 | 1/3 | 1/3 | 2/4 | 0/3 | 1/4
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 1/1 | 3/3 | 3/3 | 4/4 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - ALM201 (N=1) | Cohort 2 - ALM201 (N=1) | Cohort 3 - ALM201 (N=1) | Cohort 4 - ALM201 (N=3) | Cohort 5 - ALM201 (N=3) | Cohort 6 - ALM201 (N=4) | Cohort 7 - ALM201 (N=3) | Cohort 8 - ALM201 (N=4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device occlusion (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal vein thrombosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - ALM201 (N=1) | Cohort 2 - ALM201 (N=1) | Cohort 3 - ALM201 (N=1) | Cohort 4 - ALM201 (N=3) | Cohort 5 - ALM201 (N=3) | Cohort 6 - ALM201 (N=4) | Cohort 7 - ALM201 (N=3) | Cohort 8 - ALM201 (N=4)
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device occlusion (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 2 | 2
Injection site bruising (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Catheter site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conduction disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal vein thrombosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated after Part 1 to re-evaluate the biomarker strategy for recruitment to Part 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2014-09-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT03427073/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT03427073/SAP_001.pdf